CLINICAL TRIAL: NCT02084758
Title: The Effects of Dietary Nitrate Supplementation on Metabolic Efficiency in Patients With COPD
Brief Title: Nitrate Supplementation in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABR-47701
Record Dates: First submitted 2014-02-17; First posted 2014-03-12 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; nitrate supplementation; metabolic efficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrate supplementation (Active Comparator): Sodium nitrate solution
  Interventions: Dietary Supplement: Nitrate supplementation; Dietary Supplement: Placebo supplementation
- Placebo supplementation (Placebo Comparator): Sodium chloride solution
  Interventions: Dietary Supplement: Nitrate supplementation; Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Nitrate supplementation — 7 days of supplementation with sodium nitrate solution
Dietary Supplement: Placebo supplementation — 7 days of supplementation with sodium chloride solution

SUMMARY:
Each subject will consume (in a randomized fashion) both the intervention beverage (nitrate solution) and the placebo, separated by a 1 wk washout period. The investigators will test the hypothesis that 7 days of dietary nitrate supplementation will improve metabolic efficiency in patients with COPD compared to the placebo.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Indication metabolic inefficiency

Exclusion Criteria:

* Sodium intake limitation
* Long-term oxygen therapy
* Severe renal impairment
* Use of medications that may interact with nitrate
* Contra-indications for performing (sub)maximal cycle ergometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in metabolic efficiency during exercise | Baseline, day 7, day 14 and day 21.
  Metabolic efficiency (degree of efficiently used energy during exercise) will be assessed during the test days before and after the two supplementation periods (active and placebo) for a total timespan of 3 weeks.

SECONDARY OUTCOMES:
Change in blood pressure during exercise | Baseline, day 7, day 14 and day 21.
  Change in blood pressure will be assessed during the test days before and after the two supplementation periods (active and placebo) for a total timespan of 3 weeks.
Change in dyspnea during exercise | Baseline, day 7, day 14 and day 21.
  Change in dyspnea will be assessed during the test days before and after the two supplementation periods (active and placebo) for a total timespan of 3 weeks.
Change in cycle endurance time during exercise. | Baseline, day 7, day 14 and day 21.
  Change in cycle endurance time will be assessed during the test days before and after the two supplementation periods (active and placebo) for a total timespan of 3 weeks.
Change in oxygen uptake (VO2 mL/min) during exercise | Baseline, day 7, day 14 and day 21
  Change in oxygen uptake will be assessed during the test days before and after the two supplementation periods (active and placebo) for a total timespan of 3 weeks.
Change in Resting Energy Expenditure (REE) | Baseline, day 7, day 14 and day 21
  Change in REE will be assessed during the test days before and after the two supplementation periods (active and placebo) for a total timespan of 3 weeks.
Change in plasma concentrations of nitrate and nitrite, glucose, insulin, lactate and free fatty acids, IFABP and cardiac troponin | Baseline, day 7, day 14 and day 21
  Change in these plasma concentrations will be assessed during the test days before and after the two supplementation periods (active and placebo) for a total timespan of 3 weeks.

OTHER OUTCOMES:
VO2max and Wmax | Baseline
height, body weight and body mass index (BMI) | Baseline
Fat free mass and fat mass | Baseline
  Fat free mass and fat mass determined by DEXA-scan
Lung function | Baseline
Physical activity | During the two supplementation periods

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Schols, Prof., Study Director — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands